CLINICAL TRIAL: NCT03860519
Title: The Use of the Propeller Health Platform to Improve Inhaled Corticosteroid (ICS) Use Among Adults With Uncontrolled Persistent Asthma (Propeller Health)
Brief Title: The Use of the Propeller Health Platform to Improve Inhaled Corticosteroid (ICS) Use Among Adults With Uncontrolled Persistent Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Giselle Mosnaim, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH17-322
Record Dates: First submitted 2018-09-26; First posted 2019-03-04 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Asthma
Keywords: asthma; uncontrolled asthma; asthma medication adherence; Propeller Health; Connected Inhaler System
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The components of the intervention unique to the treatment group include: 1) access to the Propeller Health Asthma App on his/her phone, which includes tracking of ICS and SABA usage; 2) receipt of NorthShore Connect physician alerts (these will be sent by the asthma nurse on behalf of the NS physician) if he/she has "poor adherence" ie missed 4 consecutive days of all of his/her controller medication dosages and their sensor has sent heartbeat to application OR "at risk" alerts if a patient transitions to a "not well controlled" or "poorly controlled" status (defined by the NHLBI guidelines); and 3) monthly phone calls with a nurse from his/her asthma doctor's office to review ICS and SABA usage reports (provided by Propeller Health on their Propeller Health dashboard).
  Interventions: Behavioral: Electronic Medication Monitors on ICS and SABA - Active Mode; Behavioral: Asthma App Tracking of ICS/SABA Usage - Active Mode; Behavioral: NorthShore Connect Real Time ICS and SABA Usage Feedback - Yes; Behavioral: Asthma Nurse Monthly Phone Calls for ICS/SABA Usage Feedback - Yes
- Control Group (Experimental): The control group will not receive access to view the contents of the Propeller Health Asthma App on his/her phone, NorthShore Connect alerts for missing ICS or overuse of SABA, or for his/her asthma doctor (the asthma nurse will be viewing this information on behalf of the asthma doctor) to view his/her ICS and SABA use on the Propeller Health dashboard until after the 3-month study has been completed.
  Interventions: Behavioral: Electronic Medication Monitors on ICS and SABA - Silent Mode; Behavioral: Asthma App Tracking of ICS/SABA Usage - Silent Mode; Behavioral: NorthShore Connect Real Time ICS and SABA Usage Feedback - No; Behavioral: Asthma Nurse Monthly Phone Calls for ICS/SABA Usage Feedback - No

INTERVENTIONS:
Behavioral: Electronic Medication Monitors on ICS and SABA - Active Mode — The patients in the intervention group will have sensors that are "active", so that these patients receive reminders about when to use their inhalers medications.
  Other Names: MDI, Diskus
  Arms: Intervention Group
Behavioral: Electronic Medication Monitors on ICS and SABA - Silent Mode — The patients in the control group will have sensors that are "silent", so that these patients do not receive reminders about when to use their inhalers medications.
  Other Names: MDI, Diskus
  Arms: Control Group
Behavioral: Asthma App Tracking of ICS/SABA Usage - Active Mode — Patients in the intervention group will have access to their medication usage information (as collected by their sensors) via their Propeller Health applications.
  Arms: Intervention Group
Behavioral: Asthma App Tracking of ICS/SABA Usage - Silent Mode — Patients in the control group will not have access to their medication usage information (as collected by their sensors) via their Propeller Health applications.
  Arms: Control Group
Behavioral: NorthShore Connect Real Time ICS and SABA Usage Feedback - Yes — Patients in the intervention will receive feedback from the Research Nurse about their medication use and asthma control status.
  Arms: Intervention Group
Behavioral: NorthShore Connect Real Time ICS and SABA Usage Feedback - No — Patients in the intervention will not receive feedback from the Research Nurse about their medication use and asthma control status.
  Arms: Control Group
Behavioral: Asthma Nurse Monthly Phone Calls for ICS/SABA Usage Feedback - Yes — Patients in the intervention group will receive monthly calls from the Research Nurse to obtain feedback information about the Propeller Health Platform.
  Arms: Intervention Group
Behavioral: Asthma Nurse Monthly Phone Calls for ICS/SABA Usage Feedback - No — Patients in the control group will not receive monthly calls from the Research Nurse to obtain feedback information about the Propeller Health Platform.
  Arms: Control Group

SUMMARY:
This is a behavioral randomized controlled trial of adults with uncontrolled persistent asthma that tests if the Propeller Health sensor, mobile application, and dashboard can improve adherence to ICS.

ELIGIBILITY:
Inclusion Criteria:

* Under the care of a staff asthma physician (i.e. pulmonologist or allergist/immunologist) at NorthShore University HealthSystem (NS)
* Have an active NorthShore Connect (patient portal) account
* Persistent uncontrolled asthma in the past 12 months
* Active prescription for daily ICS medication for asthma

Exclusion Criteria:

* candidate refusal
* the presence of other co-morbidities (e.g. severe psychiatric disorder) that could interfere with study participation

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Short Acting Bronchodilator Medication use in Group with Propeller Health Platform Digital Technology Turned On vs Group with Propeller Health Platform Digital Technology Turned Off | 3.5 months
  Use of the Propeller Health Platform in the treatment group in active mode, compared to the attention control group in silent mode, will demonstrate a 20% change in SABA use and/or minimal clinically important difference (three points) change on the ACT and/or change from ACT score ≤ 19 to ≥20, at 3-months. The 20% change in SABA use = 20 point change (e.g. if a participants uses SABA 40% of days over the 2 week run-in period, and they change SABA use to 20% of days during the final 14 days of the active treatment period, that will equal a 20 point change. If SABA use changes from 40% of days over the 2- week run-in period to 32% of days during the final 14 days of the active treatment period, this will not be considered a 20 point change).

SECONDARY OUTCOMES:
Participant and clinician satisfaction as assessed by brief post-study survey of Propeller Health Platform Digital Technology | 3.5 months
  Study staff developed a brief survey using open-ended questions (i.e. 20 questions, no scales used, no minimum or maximum scores are applicable) to ask participants and clinicians whether they were satisfied using the Propeller Health Platform Digital Technology. Standardized instruments are not being used.
Inhaled Corticosteroid Medication taking Behavior in the Group using Propeller Health Platform Digital Technology Turned On vs Group using Propeller Health Platform Digital Technology Turned Off | 3 months
  To determine if two Propeller Health Platform Digital Technology arms (i.e. Arm #1= Technology in active "on" mode and Arm #2= Technology in passive "off" mode) demonstrate a change in inhaled corticosteroid medication taking behavior at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Mosnaim, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

REFERENCES:
- [Derived] Mosnaim GS, Stempel DA, Gonzalez C, Adams B, BenIsrael-Olive N, Gondalia R, Kaye L, Shalowitz M, Szefler S. Electronic medication monitoring versus self-reported use of inhaled corticosteroids and short-acting beta2-agonists in uncontrolled asthma. J Asthma. 2022 Oct;59(10):2024-2027. doi: 10.1080/02770903.2021.1996600. Epub 2021 Nov 2. PMID 34699302
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Application+of+Human+Augmentics%3A+A+Persuasive+Asthma+Inhaler
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/25609351
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+Impact+of+Peer+Support+and+mp3+Messaging+on+Adherence+to+Inhaled+Corticosteroids+in+Minority+Adolescents+with+Asthma%3A+A+Randomized+Controlled+Trial